CLINICAL TRIAL: NCT00331838
Title: A Multicenter, Randomized, Double-Blind, Double-Dummy, Parallel Group, Dose Response Study of Subcutaneous AVE5026 With an Enoxaparin Calibrator Arm in the Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Knee Replacement Surgery
Brief Title: Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Knee Replacement Surgery
Acronym: TREK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DRI6243; 2005-006202-26 (EudraCT Number)
Record Dates: First submitted 2006-05-18; First posted 2006-05-31 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Venous Thromboembolism
Keywords: Prevention; Venous Thrombosis; Orthopedic Surgery
MeSH Terms: conditions — Venous Thromboembolism; Venous Thrombosis | interventions — AVE 5026; enoxaparin sodium; Enoxaparin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Semuloparin 5 mg (Experimental): Semuloparin sodium 5 mg + Placebo (for Enoxaparin sodium) once daily for 4-10 days with an initial dose given 12 hours before or 8 hours after surgery depending on the willingness of the investigator
  Interventions: Drug: Semuloparin sodium; Drug: Placebo (for Enoxaparin sodium)
- Semuloparin 10 mg (Experimental): Semuloparin sodium 10 mg + Placebo (for Enoxaparin sodium) once daily for 4-10 days with an initial dose given 12 hours before or 8 hours after surgery depending on the willingness of the investigator
  Interventions: Drug: Semuloparin sodium; Drug: Placebo (for Enoxaparin sodium)
- Semuloparin 20 mg (Experimental): Semuloparin sodium 20 mg + Placebo (for Enoxaparin sodium) once daily for 4-10 days with an initial dose given 12 hours before or 8 hours after surgery depending on the willingness of the investigator
  Interventions: Drug: Semuloparin sodium; Drug: Placebo (for Enoxaparin sodium)
- Semuloparin 40 mg (Experimental): Semuloparin sodium 40 mg + Placebo (for Enoxaparin sodium) once daily for 4-10 days with an initial dose given 12 hours before or 8 hours after surgery depending on the willingness of the investigator
  Interventions: Drug: Semuloparin sodium; Drug: Placebo (for Enoxaparin sodium)
- Semuloparin 60 mg (Experimental): Semuloparin sodium 60 mg + Placebo (for Enoxaparin sodium) once daily for 4-10 days with an initial dose given 12 hours before or 8 hours after surgery depending on the willingness of the investigator
  Interventions: Drug: Semuloparin sodium; Drug: Placebo (for Enoxaparin sodium)
- Enoxaparin 40 mg (Active Comparator): Enoxaparin sodium 40 mg + Placebo (for Semuloparin sodium) once daily for 4-10 days with an initial dose given 12 hours before or 8 hours after surgery depending on the willingness of the investigator
  Interventions: Drug: Enoxaparin sodium; Drug: Placebo (for Semuloparin sodium)
- Placebo pre-op / Semuloparin 20 mg (Experimental): Placebo (for Semuloparin sodium) + Placebo (for Enoxaparin sodium) 12 hours before surgery then,
  Semuloparin sodium 20 mg + Placebo (for Enoxaparin sodium) once daily for 4-10 days with an initial dose given 8 hours after surgery
  Interventions: Drug: Semuloparin sodium; Drug: Placebo (for Enoxaparin sodium); Drug: Placebo (for Semuloparin sodium)
- Placebo pre-op / Semuloparin 40 mg (Experimental): Placebo (for Semuloparin sodium) + Placebo (for Enoxaparin sodium) 12 hours before surgery then,
  Semuloparin sodium 40 mg + Placebo (for Enoxaparin sodium) once daily for 4-10 days with an initial dose given 8 hours after surgery
  Interventions: Drug: Semuloparin sodium; Drug: Placebo (for Enoxaparin sodium); Drug: Placebo (for Semuloparin sodium)

INTERVENTIONS:
Drug: Semuloparin sodium — 0.8 mL solution in Type I amber glass vials
  Subcutaneous injection
  Other Names: AVE5026
  Arms: Placebo pre-op / Semuloparin 20 mg; Placebo pre-op / Semuloparin 40 mg; Semuloparin 10 mg; Semuloparin 20 mg; Semuloparin 40 mg; Semuloparin 5 mg; Semuloparin 60 mg
Drug: Placebo (for Enoxaparin sodium) — 0.4 mL solution in ready-to-use prefilled syringe strictly identical in appearance containing the same volume but without active component
  Subcutaneous injection
  Arms: Placebo pre-op / Semuloparin 20 mg; Placebo pre-op / Semuloparin 40 mg; Semuloparin 10 mg; Semuloparin 20 mg; Semuloparin 40 mg; Semuloparin 5 mg; Semuloparin 60 mg
Drug: Enoxaparin sodium — 0.4 mL solution in ready-to-use pre-filled syringe
  Subcutaneous injection
  Other Names: Lovenox®
  Arms: Enoxaparin 40 mg
Drug: Placebo (for Semuloparin sodium) — 0.8 ml solution in type I amber glass vials strictly identical in appearance containing the same volume but without active component
  Subcutaneous injection
  Arms: Enoxaparin 40 mg; Placebo pre-op / Semuloparin 20 mg; Placebo pre-op / Semuloparin 40 mg

SUMMARY:
The primary objective was to demonstrate the dose-response of Semuloparin sodium (AVE5026) for the prevention of Venous Thromboembolism [VTE] in patients undergoing total knee replacement [TKR] surgery.

Secondary objectives were to evaluate the safety (incidence of major bleeding) of AVE5026, to document the efficacy and safety of AVE5026 post-operative regimens, and to assess the pharmacokinetic parameters of AVE5026.

DETAILED DESCRIPTION:
The randomization had to take place before the first study drug injection.

The total duration of observation per participant was 27-33 days from surgery broken down as follows:

* 4 to 10-day double-blind treatment period;
* Follow-up period up to Day 30 ± 3 after surgery.

Mandatory bilateral venography of the lower limbs had to be performed between 5 to 11 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled to undergo elective total knee replacement or revision of a primary procedure performed ≥ 6 months prior to study entry.

Exclusion Criteria:

* Any major orthopedic surgery in the 3 months prior to study entry;
* Clinical signs or symptoms of DVT or PE within the last 12 months or known post-phlebitic syndrome;
* Known sensitivity to iodine or contrast dyes;
* Recent stroke or myocardial infarction;
* High risk of bleeding;
* Treatment with other anti-thrombotic agents within 7 days prior to surgery;
* Any contra-indication to Unfractionated Heparin or Low Molecular Weight Heparin;
* Pregnant or nursing woman, or woman of childbearing potential who is not using an effective contraceptive method.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 705 (Actual)
Dates: Start 2006-05; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Venous Thromboembolism Event (VTE) or VTE-related Death | From surgery to Day 11 or the day of mandatory venography, whichever came first
  VTE included any Deep Vein Thrombosis [DVT] identified on mandatory venography of the lower limbs; symptomatic DVT and/or non-fatal pulmonary embolism [PE] before mandatory examination; VTE related deaths included fatal PE or deaths which could not be attributed to a documented cause and for which PE could not be ruled out. All events were to be confirmed by a Central Independent Adjudication Committee [CIAC] based on venographies, scheduled or unscheduled, and other available diagnostic tests (ultrasonography, ventilation/perfusion lung scan, pulmonary angiography, autopsy report, etc).

SECONDARY OUTCOMES:
Number of Participants Who Experienced DVT | From surgery up to Day 11 or the day of mandatory venography, whichever came first
Number of Participants Who Experienced Symptomatic VTE | From surgery up to Day 11 or the day of mandatory venography, whichever came first
  Symptomatic VTE included:
  * suspected DVT confirmed by the CIAC based on compression ultrasonography or venography;
  * suspected PE confirmed by the CIAC based on perfusion/ventilation lung scan, pulmonary angiography or spiral computerized tomography.
Number of Participants Who Experienced Bleedings | From 1st study drug injection up to 3 days after last study drug injection (median duration of approximately 11 days)
  Bleedings were centrally and blindly reviewed by the CIAC and classified as:
  * "Major" (fatal bleeding, bleeding that was retroperitoneal or intracranial or that involved any other critical organ (e.g. eye, adrenal gland, pericardium or spine), surgical site bleeding leading to intervention, non-surgical site bleeding requiring surgical intervention or with a bleeding index ≥2);
  * "Minor" (overt bleeding considered more than expected but not meeting the criteria for major bleeding);
  * "Criteria for bleeding event not satisfied" (not meeting the criteria for major or minor bleeding).
Number of Participants Who Required Initiation of Curative Anticoagulant or Thrombolytic Treatment After VTE Assessment | From surgery up to Day 11 or the day of mandatory venography, whichever came first
  Initiation of curative anticoagulant or thrombolytic treatment after VTE assessment was defined from investigator's answers to questions asked after diagnostic tests for suspected VTE and/or the mandatory venography.

OTHER OUTCOMES:
Number of Deaths | From 1st study drug injection up to 3 days after last study drug injection (median duration of approximately 11 days)
  All deaths were centrally and blindly reviewed by the CIAC and classified as "Fatal PE", "PE not excluded", "Fatal bleeding" and "Death not associated with VTE or bleeding" based on relevant documentation (e.g. autopsy report).
Platelets Count: Number of Participants With Potentially Clinically Significant Abnormalities [PCSA] | From 1st study drug injection up to 3 days after last study drug injection (median duration of approximately 11 days)
  PCSA are abnormal values considered medically important by the Sponsor according to predefined criteria based on literature review. Threshold for platelet counts was defined as <100 Giga/L.
Liver Function: Number of Participants With Potentially Clinically Significant Abnormalities [PCSA] | From 1st study drug injection up to 3 days after last study drug injection (median duration of approximately 11 days)
  Thresholds were defined as follows:
  * Alanine Aminotransferase [ALAT] >3 Upper Normal Limit [ULN];
  * Total Bilirubin [TB] ≥34 μmol/L;
  * ALAT ≥3 ULN and TB ≥34 μmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Michael LASSEN, MD, Study Chair — Hoersholm Hospital (Denmark)
Locations (19):
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Santiago, Chile
- Sanofi-Aventis Administrative Office, Bogotá, Colombia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, México, Mexico
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Makati City, Philippines
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Bangkok, Thailand
- Sanofi-Aventis Administrative Office, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Lassen MR, Dahl OE, Mismetti P, Destree D, Turpie AG. AVE5026, a new hemisynthetic ultra-low-molecular-weight heparin for the prevention of venous thromboembolism in patients after total knee replacement surgery--TREK: a dose-ranging study. J Thromb Haemost. 2009 Apr;7(4):566-72. doi: 10.1111/j.1538-7836.2009.03301.x. Epub 2009 Jan 24. PMID 19187076